CLINICAL TRIAL: NCT05112692
Title: Progestin-primed Ovarian Stimulation Protocol Versus GnRH Antagonist Protocol in Polycystic Ovary Syndrome Patients Undergoing IVF/ICSI Cycles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PPOS in ICSI for PCOS
Record Dates: First submitted 2021-10-04; First posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-10

CONDITIONS: PCOS (Polycystic Ovary Syndrome) of Bilateral Ovaries
Keywords: Progestin; ICSI; antagonist
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Dydrogesterone; cetrorelix; Menotropins; Triptorelin Pamoate; Chorionic Gonadotropin; Cryopreservation; Estradiol; Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PPOS group (Active Comparator): Patients will be coadministered with Human Menopausal Gonadotrophin (HMG) 150-225 international unit/day (IU/d) via intramuscular injection and oral DYG 20mg/d from menstrual cycle day 3 (MC3) to the day of triggering. The starting dose of HMG is 150IU/day for patients with a high antral follicle count >20 or slightly elevated basal FSH (7-10IU/L), and a daily dose of 225IU HMG is used for the other patients. The dose will be adjusted after day 5 of stimulation based on the ovarian response as assessed by serum hormone levels and transvaginal ultrasonography
  Interventions: Drug: Dydrogesterone Tablets; Drug: human menopausal gonadotropin; Drug: triptorelin 0.1 mg; Drug: human chorionic gonadotropin; Procedure: cryopreservation; Drug: Estradiol Valerate and progesterone
- GnRH antagonist (Active Comparator): In the fixed GnRH antagonist protocol, daily s.c. administration of Cetrotide 0.25 mg will be initiated at 6th day of stimulation. HMG (150-225IU) will be administered daily from menstrual cycle day 3, and follicular monitoring will be performed every 2 to 3 days after 5 days of injections. The dose of hMG will be adjusted according to the ovarian response, as monitored by ultrasonography and the measurement of serum sex steroids. Treatment with hMG and GnRH antagonist will continue daily until the day when final oocyte maturation is triggered
  Interventions: Drug: cetrorelix 0.25mg; Drug: human menopausal gonadotropin; Drug: triptorelin 0.1 mg; Drug: human chorionic gonadotropin; Procedure: cryopreservation; Drug: Estradiol Valerate and progesterone

INTERVENTIONS:
Drug: Dydrogesterone Tablets — first arm will be coadministered gonadotrophins with 20mg dydrogesterone till day of trigger second arm will be subjected to fixed GnRH antagonist protocol then will do Freeze All in both arms then frozen embryo transfer next cycle
  Arms: PPOS group
Drug: cetrorelix 0.25mg — In the fixed GnRH antagonist protocol, daily s.c. administration of Cetrotide 0.25 mg will be initiated at 6th day of stimulation. HMG (150-225IU) will be administered daily from menstrual cycle day 3.
  Arms: GnRH antagonist
Drug: human menopausal gonadotropin — (150-225IU) will be administered daily from menstrual cycle day 3 till day ot trigger
Drug: triptorelin 0.1 mg — When the dominant follicles reach a diameter of 18mm, the final stage of oocyte maturation will be induced with injections of 100µg of triptorelin s.c combined with 1000IU of hCG i.m
Drug: human chorionic gonadotropin — When the dominant follicles reach a diameter of 18mm, the final stage of oocyte maturation will be induced with injections of 100µg of triptorelin s.c combined with 1000IU of hCG i.m
Procedure: cryopreservation — All of the follicles greater than 10mm in diameter will be aspirated. The oocytes are inseminated approximately 4-6hours after follicular aspiration by a conventional IVF method or intracytoplasmic sperm injection, based on the sperm quality On day 3, high quality embryos are cryopreserved by means of vitrification
Drug: Estradiol Valerate and progesterone — Endometrium will be prepared using step-up oral estrogen protocols. On day 14 of estrogen administration, endometrial thickness will be assessed and serum progesterone level will be measured, with cycles to be cancelled according to the arbitrary thresholds of 7.0 mm and 1.5 ng/mL, respectively. Progesterone administration will be started on the morning (am) of day 15, with the start date of progesterone and the day of blastocyst cryopreservation used to coordinate the day of FET

SUMMARY:
The purpose of this trial is to compare the efficacy and safety of the PPOS protocol to the GnRH antagonist protocol in patients with PCOS who are undergoing IVF/ICSI cycles.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is a common metabolic dysfunction and heterogeneous endocrine disorder. It is the most common cause of anovulatory infertility, affecting approximately 10%-18% of reproductive age women worldwide.

It is usually characterized by a clustering of hyperandrogenism, hypersecretion of luteinizing hormone (LH) and hyperinsulinaemia, which could result in the arrest of ovarian follicular growth, oligo-ovulation or anovulation, menstrual dysfunction, hirsutism, infertility, pregnancy and/or neonatal complications.

Women with PCOS undergoing IVF or Intracytoplasmic sperm injection (ICSI) treatment because of infertility are increasing in number, and these patients have been well described, typically characterized by producing an increased number of oocytes but are often of poor quality leading to lower fertilization, implantation, and pregnancy rates and a higher miscarriage rate and incidence of ovarian hyperstimulation syndrome.

Increasing evidence raises the issue that impaired oocyte maturation and developmental competence in women with PCOS are possibly linked to abnormal endocrine/ paracrine factors, metabolic dysfunction and alterations in the intrafollicular microenvironment during folliculogenesis and follicle maturation.

Several clinical ovarian stimulation protocols have been used so far in women with PCOS undergoing IVF treatment to prevent a premature LH surge during controlled ovarian stimulation (COS); these primarily include gonadotropin-releasing hormone (GnRH) agonist or antagonist protocols.

GnRH antagonists can competitively inhibit endogenous GnRH and produce an immediate and rapid decline in LH and Follicle-stimulating hormone (FSH) levels without the flare effect of a GnRH agonist, and their administration by subcutaneous injection in the late follicular phase prevents an LH surge.

With progress in embryo vitrification techniques, many studies have suggested that pregnancies that arise from the transfer of frozen-thawed IVF embryos appear to have better perinatal and pregnancy outcomes. Thus, GnRH antagonist regimens combined with a freeze-all strategy for women with PCOS are currently accepted as the most routine IVF procedures.

The progesterone's pituitary suppression was recently used in controlled ovarian stimulation and approved its efficacy in terms of low incidence of premature LH surge and comparable pregnancy outcomes to short protocols in infertile women of normal ovarian reserve and polycystic ovarian syndrome.

These data indicated that progestin treatment might improve oocyte quality compared with a GnRH antagonist during COS in these patients, plus there were the advantages of an oral administration route instead of repeated injections of GnRH antagonist, a lower drug price and more control over LH levels, which can reduce the patients' discomfort and costs.

Furthermore, to avoid a low response of the hypothalamic pituitary ovarian axis, a double trigger with GnRHa and a low dose of Human chorionic gonadotropin (hCG)(1000IU) was used to induce final oocyte maturation without increasing the risk of moderate or severe Ovarian hyperstimulation syndrome (OHSS).

Choosing the appropriate progestin is crucial to the success of the Progestin-primed ovarian stimulation protocol (PPOS). Previous studies have shown that both Medroxyprogesterone acetate (MPA) and Utrogestan are effective oral alternatives for the PPOS protocol.

MPA is preferred over Utrogestan because the administration of a natural exogenous progesterone, such as Utrogestan, can interfere with serum progesterone measurement and lead to the neglect of possible premature luteinization. However, the use of MPA during ovarian stimulation may lead to stronger pituitary suppression and thus may require a higher dosage of gonadotrophin and a longer ovarian stimulation duration than that of the conventional ovarian stimulation protocol. Therefore, the investigators need to test more synthetic progestins to find the most suitable option for PPOS.

Dydrogesterone (DYG), which has a molecular structure similar to that of natural progesterone, is widely used for hormone replacement therapy, endometriosis treatment, menstrual disorders and luteal support in pregnancy and threatened miscarriage. However, unlike MPA, the use of DYG under the recommended dosage (10-20 mg) does not inhibit ovulation, and thus, the use of DYG as an alternative to MPA and as an appropriate progestin in the PPOS regimen has yet to be explored.

In this study, the investigators hypothesize that DYG can be used as an alternative progestin in the PPOS protocol. A randomized controlled trial (RCT) is designed to investigate cycle characteristics and endocrinological profiles of patients taking gonadotrophin while using DYG co-treatment, and to compare pregnancy outcomes in first frozen embryo transfer (FET) cycles with GNRH antagonist protocol as a control.

ELIGIBILITY:
Inclusion Criteria:

* Women who have a history of infertility ≥1year.
* Ages between 20 and 35 years.
* Patients diagnosed with PCOS according to the revised 2003 Rotterdam consensus and met 2 out of 3 criteria as follows (Rotterdam, 2004):

  * Oligo- and/or anovulation.
  * Biochemical and/or clinical evidence of hyperandrogenism.
  * Polycystic ovarian morphology on ultrasound (the presence of ≥12 antral follicles (≤9mm) and/or ovarian volume >10mL on transvaginal ultrasonographic scanning).

Other etiologies of hyperandrogenism and ovulatory dysfunction will be excluded, including androgen-secreting tumors, congenital adrenal hyperplasia, hyperprolactinemia and thyroid disease.

Exclusion Criteria:

* Endometriosis grade 3 or higher.
* Documented ovarian failure, including basal FSH above 10IU/L.
* Clinically significant systemic disease, or other endocrine disorders, including 21-hydroxylase deficiency, uncorrected thyroid disease or suspected Cushing's syndrome.
* Patients who in the previous 3 months received hormonal treatments or other medications known to affect reproductive function, including oral contraceptives and GnRH agonists.
* Documented history of ovarian surgery including laparoscopic ovarian drilling, ovarian endometrioma stripping and unilateral oophorectomy
* Previous diagnosis of congenital (septate uterus, duplex uterus, uterus bicornis and uterus unicornis) or acquired (intrauterine adhesion, submucosal myomas and adenomyosis) uterine anomalies
* History of recurrent spontaneous abortion, defined as three or more previous spontaneous pregnancy losses
* Abnormal chromosomal karyotype in either of the partners.
* Inability to comply with the study procedures.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate | 6 weeks after embryo transfer
  clinical pregnancy is defined as presence of gestational sac on ultrasound performed at 6 weeks after ET. A clinical pregnancy rate is defined as number of clinical pregnancies divided by number of ET procedures.

SECONDARY OUTCOMES:
the incidence of premature LH surges | trigger day
  premature LH surge is increased serum LH more than twice the baseline or more than 15 Milli-international units per milli litre
fertilization rate | baseline
  number of embryos formed per 100 injected oocytes
implantation rate | baseline
  number of gestational sacs per 100 transferred embryos
ongoing pregnancy rate | baseline
  number of viable pregnancies beyond 8-10 weeks of gestation
live birth rate | baseline
  delivery of any viable infant at 28 weeks or longer gestation after embryo transfer